CLINICAL TRIAL: NCT01095419
Title: Effects of Massage Therapy on Sleep Quality After Coronary Artery Bypass Graft Surgery
Brief Title: Effects of Massage Therapy on Sleep After Heart Surgery
Acronym: MT and CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação Zerbini (Unknown)
Responsible Party: Effects of Massage Therapy on Sleep Quality after Coronary Artery Bypass Graft Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-CABG
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: massage therapy; sleep quality; coronary artery bypass grafting surgery; Patients after Coronary Artery Bypass Graft Surgery
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients were seated in a chair for the same period then those from MT group, but did not receive intervention
  Interventions: Other: Control
- Massage Therapy (Experimental): Patients in the postoperative period of coronary artery bypass graft surgery, which receive intervention for 3 consecutive days
  Interventions: Other: Massage Therapy

INTERVENTIONS:
Other: Massage Therapy — After discharge from the intensive care unit to the ward during the postoperative period, patients which were randomized for 3 nights to receive intervention (Massage Therapy)which were consisted of massage of the neck, shoulders, and back. The massage was initiated with light manual compression and progressed to deep compression. The compression was performed with the inner region of the fingers, hand-shaped clamp, and friction (digital compression with the thumb) on trigger points, cervical traction, and mobilization in all planes (front, back, and sides)
  Arms: Massage Therapy
Other: Control — no intervention
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of Massage Therapy for improving the quality of sleep in patients on postoperative period of coronary artery bypass graft surgery (CABG).

DETAILED DESCRIPTION:
Patients We evaluated patients admitted to the ward waiting for elective CABG surgery.

Preoperative evaluation The preoperative clinical assessment consisted of obtaining information regarding demographics and personal characteristics.

Postoperative protocol and evaluation After discharge from the intensive care unit to the ward during the postoperative period, the patients were randomized to 3 nights of sitting for 10 minutes, with no intervention (Control) or to MT. Briefly, MT consisted of massage of the neck, shoulders, and back. The massage was initiated with light manual compression and progressed to deep compression. The compression was performed with the inner region of the fingers, hand-shaped clamp, and friction (digital compression with the thumb) on trigger points, cervical traction, and mobilization in all planes (front, back, and sides). The massage was finished with light manual compression. During the study period, all patients completed a sleep diary containing the time they went to sleep, woke up, and took daytime naps. The patients completed a VAS for pain and fatigue (similar to the preoperative evaluation described previously) as well as a VAS for sleep on days 1, 2, and 3, corresponding to the morning following the intervention that was performed on the previous night.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included patients of both genders, between 40 to 80 years of age which were waiting for Coronary artery bypass graft surgery.

Exclusion Criteria:

* Patients with body mass index (BMI) ≥35kg/m2
* Regular alcohol consumption
* Chronic use of hypnotics
* A previous diagnosis of sleep disorders
* Previous surgeries performed in the last 24 months
* The inability to read and write. We also excluded patients who underwent valve surgery combined with CABG, the presence of a thoracic drain, and ICU stay longer than 5 days in the postoperative period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Effects of Massage Therapy on quality of sleep | 3 days after return to the ward

SECONDARY OUTCOMES:
Effect of massage therapy on pain and fatigue complaints | 3 days after return to the ward

CONTACTS AND LOCATIONS:
Overall Officials: Flávia B. Nerbass, PT, Principal Investigator — University of Sao Paulo; Geraldo Lorenzi-Filho, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- Heart Institute -University of São Paulo School of Medicine, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nerbass FB, Feltrim MI, Souza SA, Ykeda DS, Lorenzi-Filho G. Effects of massage therapy on sleep quality after coronary artery bypass graft surgery. Clinics (Sao Paulo). 2010;65(11):1105-10. doi: 10.1590/s1807-59322010001100008. PMID 21243280